CLINICAL TRIAL: NCT00126295
Title: Evaluation of a Computer-Generated Individualised Written Education Package for Patients Following Stroke and Their Carers
Brief Title: Evaluation of an Individualised Written Education Package for Stroke Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Benefits Fund of Australia (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: 2002000023
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2005-08-19 (Estimated); Status verified 2005-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Device: 'What you need to know about stroke' education package

SUMMARY:
The primary aim of the randomised controlled trial was to evaluate the effectiveness of a tailored written education package ("What you need to know about stroke") on the outcomes of:

* Knowledge about stroke, self-efficacy, anxiety, depression, perceived health status, satisfaction with the content and presentation of the information received, and desire for additional information for patients following stroke and
* Knowledge about stroke, self-efficacy, anxiety, depression, satisfaction with the content and presentation of the information received, and desire for additional information for their carers.

A secondary aim was to evaluate the effect of written information on the outcomes of knowledge about stroke, self-efficacy, anxiety, depression, and perceived health status of patients following stroke and on knowledge about stroke, self-efficacy, anxiety, and depression of their carers.

ELIGIBILITY:
Inclusion Criteria:

* Had a stroke or transient ischemic attack (TIA) or was the informal carer of a person who had a stroke or TIA;
* Had a reported English-proficiency level, corrected hearing and vision, and communication status adequate to participate in an interview and complete assessment tasks;
* Did not have reported or observable dementia;
* Lived within 50km of the hospital, for ease of follow-up; and
* Was medically stable.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 2003-06; Study Completion 2005-05

PRIMARY OUTCOMES:
knowledge about stroke
self-efficacy
anxiety
depression
perceived health status (patients only)
satisfaction with the content and presentation of the information received
desire for additional information

CONTACTS AND LOCATIONS:
Overall Officials: Tammy C Hoffmann, Principal Investigator — The University of Queensland; Kryss McKenna, Principal Investigator — The University of Queensland; Linda Worrall, Principal Investigator — The University of Queensland; Stephen Read, Principal Investigator — Royal Brisbane Hospital
Locations (1):
- Royal Brisbane Hospital, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082